CLINICAL TRIAL: NCT06944795
Title: A Short Wave Infrared Otoscope for Objective Middle Ear Effusion Diagnosis
Brief Title: SWIR Otoscopy Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Tulio Valdez, Professor of Otolaryngology - Head & Neck Surgery, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB 44549; R01DC021326 (NIH)
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Otitis Media; Otitis Media Chronic; Otitis Media Effusion
Keywords: middle ear infections; ear infections; pediatric ear infections; otitis media; chronic otitis media; chronic otitis media with effusion
MeSH Terms: conditions — Otitis Media; Otitis Media with Effusion; Otitis

STUDY DESIGN:
Masking Description: The physician who performs the tympanostomy tube placement procedure will not be analyzing the SWIR otoscope images. A different physician and a computer program will analyze the images for presence or absence of fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SWIR otoscope + white light otoscope (Experimental): Patients who are undergoing a tympanostomy tube placement as part of standard of care will have their middle ears imaged with the SWIR otoscope. The SWIR otoscope will record images/recordings of the SWIR otoscope and the white light otoscope, therefore, there will only be one arm of the study because all patients will be imaged with the white light and the SWIR.
  Interventions: Device: SWIR device

INTERVENTIONS:
Device: SWIR device — A Short Wave Infrared (SWIR) Otoscope will record images for both the SWIR and white light video otoscopes. These images of the middle ear will be recorded in AVI format.

SUMMARY:
The aim of this study is to provide preliminary data to support future studies to demonstrate that the short wave infrared (SWIR) otoscope is a better diagnostic tool than a white light otoscope for diagnosing middle ear infections (otitis media). Patients who are having a tympanostomy tube placement procedure will be participating in this study. Imaging will be performed with the white light otoscope and the SWIR otoscope to determine presence of absence of fluid. The SWIR otoscope will gather SWIR data and white light data simultaneously. As part of standard of care, patients who come in for this procedure have removal of middle ear fluid as part of their procedure, which will confirm presence or absence of fluid.

DETAILED DESCRIPTION:
Millions of children worldwide obtain an antibiotic prescription for treatment of an ear infection (otitis media), and this has been ranked in the top five conditions for direct medical spending for those under 18 years of age. Otitis media is responsible for the vast majority of tympanostomy tube placements, the most common surgical procedure in the US in children with over 600,000 cases per year. Otitis media is inadequately diagnosed and consequently mistreated. Diagnosis is estimated at 51% for US pediatricians, with over-diagnosis occurring 26% of the time. Accurate diagnosis of otitis media can be an issue as it requires a physician to differentiate between various forms of middle ear conditions. The standard of care (SOC) for diagnosing otitis media is pneumotoscopy by eye or using a white light video otoscope. This technique has advantages, but it suffers from subjective interpretations, especially in the hands of inexperienced practitioners. Our team developed the first otoscope sensitive to short wave infrared (SWIR) light for objective identification of middle ear effusions. The SWIR otoscope collects both the information normally seen by a white light otoscope, and SWIR light. The goal with this research is to evaluate the SWIR otoscope against the white light otoscope currently used as the standard of care diagnostic tool in clinic settings. Patients who are undergoing a tympanostomy tube placement procedure will be eligible for this study. In the operating room, imaging will be performed with the SWIR otoscope, which will gather images of both SWIR data and white light data simultaneously. As part of SOC, patients who come into the operating room for the procedure will have removal of middle ear fluid as part of the procedure. The physician performing the procedure will take note of the presence or absence of middle ear fluid. A different physician and a computer program will analyze the images of the SWIR otoscope for presence or absence of middle ear fluid in the image. These results will be compared with the notes taken during the procedure regarding presence or absence of ear fluid.

ELIGIBILITY:
Inclusion Criteria:

* Ages 1-17
* Being seen in the Ear, Nose, and Throat Clinic at Lucile Packard Childrens Hospital
* Undergoing tympanostomy tube placement as part of standard of care
* Parents and/or patient has the ability to understand and the willingness to sign a written informed consent form or assent form.

Exclusion Criteria:

* Patients under 1 year of age or 18 and older
* Participants not meeting the inclusion criteria

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of accurate diagnoses made by SWIR otoscope as confirmed by presence/absence of fluid during tympanostomy tube placement | 30 minutes
  Patients who are having a tympanostomy tube placement procedure at the LPCH will undergo removal of middle ear fluid as part of their standard of care. During the procedure, the physician will use the SWIR otoscope to take images using the SWIR and the white light otoscope. The physician conducting the procedure will take note of whether there was a presence of absence of middle ear fluid. A different physician and a computer program. The accuracy of the otscopes will be determined by comparing the physician and program's diagnoses to physical presence of fluid when the ear is drained during the tympanostomy tube placement.

CONTACTS AND LOCATIONS:
Overall Officials: Tulio Valdez, MD, MSc, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - Children's National Hospital, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martynkina LP, Vengerov IuIu, Bespalova IA, Sergeeva GI, Tikhonenko AS. [Structure of the interphase chromatin in the ciliata Bursaria truncatella macronucleus. II. Loop organization of inactive chromatin clumps]. Mol Biol (Mosk). 1984 Jan-Feb;18(1):272-6. Russian. PMID 6423968
- [Background] Kashani RG, Mlynczak MC, Zarabanda D, Solis-Pazmino P, Huland DM, Ahmad IN, Singh SP, Valdez TA. Shortwave infrared otoscopy for diagnosis of middle ear effusions: a machine-learning-based approach. Sci Rep. 2021 Jun 15;11(1):12509. doi: 10.1038/s41598-021-91736-9. PMID 34131163
- [Background] Pichichero ME. Diagnostic accuracy, tympanocentesis training performance, and antibiotic selection by pediatric residents in management of otitis media. Pediatrics. 2002 Dec;110(6):1064-70. doi: 10.1542/peds.110.6.1064. PMID 12456901
- [Background] Pichichero ME, Poole MD. Assessing diagnostic accuracy and tympanocentesis skills in the management of otitis media. Arch Pediatr Adolesc Med. 2001 Oct;155(10):1137-42. doi: 10.1001/archpedi.155.10.1137. PMID 11576009
- [Background] Coker TR, Chan LS, Newberry SJ, Limbos MA, Suttorp MJ, Shekelle PG, Takata GS. Diagnosis, microbial epidemiology, and antibiotic treatment of acute otitis media in children: a systematic review. JAMA. 2010 Nov 17;304(19):2161-9. doi: 10.1001/jama.2010.1651. PMID 21081729
- [Background] Grubb MS, Spaugh DC. Treatment failure, recurrence, and antibiotic prescription rates for different acute otitis media treatment methods. Clin Pediatr (Phila). 2010 Oct;49(10):970-5. doi: 10.1177/0009922810370363. Epub 2010 Jun 3. PMID 20522607